CLINICAL TRIAL: NCT06211647
Title: A Clinical Study to Evaluate the Safety, Tolerability, Dosimetry and Preliminary Efficacy of [177Lu]Lu-XT117 Injection in FAP-positive Patients With Advanced Solid Tumors
Brief Title: A Clinical Study of [177Lu]Lu-XT117 Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruimin Wang (Other)
Collaborators: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor-Investigator, Ruimin Wang, Chief of Nuclear Medicine Department, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT-XTR017-1-01 V1.1
Record Dates: First submitted 2023-12-20; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [177Lu]Lu-XT117 dose escalation (Experimental)
  Interventions: Drug: [177Lu]Lu-XT117

INTERVENTIONS:
Drug: [177Lu]Lu-XT117 — [177Lu]Lu-XT117 is a radiopharmaceutical therapy in which an beta emitter, Lu-177, is conjugated to XT117. Patients will receive [177Lu]Lu-XT117 administration at fixed dose levels at an interval of 6 weeks between each dose.

SUMMARY:
This is a single-center, single-arm clinical study to evaluate the safety, tolerability, dosimetry and preliminary efficacy of [177Lu]Lu-XT117 injection in patients with FAP-positive advanced solid tumors. Dose escalation will be conducted to determine the Dose Limiting Toxicity (DLT), Maximum Tolerated Dose (MTD), Recommended Phase 2 Dose (RP2D), and to assess dosimetry characteristics.

ELIGIBILITY:
Key Inclusion Criteria:

* ≥18 years old
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 to 1
* Confirmed as malignant solid tumor by histopathology
* Have measurable lesions based on RECIST 1.1
* Have failed standard treatment (disease progression or intolerance) or lack of standard treatment
* Positive FAP expression confirmed by FAP PET/CT
* Sufficient bone marrow capacity and organ function

Key Exclusion Criteria:

* High intensity and large amounts of off-target uptake detected by FAP molecular imaging, and were assessed as inappropriate for [177Lu]Lu-XT117 therapy by the investigators
* Previous systemic antitumor therapy (including prior chemotherapy, radiotherapy, immunotherapy, and other investigational drugs) ≤28 days before receiving study therapy; previous treatment with Chinese medicine with anti-tumor indications within 2 weeks before receiving study therapy
* Uncontrolled diabetes, with baseline fasting blood glucose > 2×ULN
* Clinically significant serious cardiovascular disease, including but not limited to: a. >Grade II congestive heart failure as per New York Heart Association (NYHA) ; b. Unstable angina pectoris or myocardial infarction within 6 months before the first administration of the study drug; c. Severe arrhythmia within 6 months prior to the first administration; d. Poorly controlled hypertension (patients who keep the blood pressure to ≤ Grade 2 hypertension [CTCAE5.0] with hypotensors are acceptable for enrollment); e. QTc>450 ms (male) or 470 ms (female), congenital prolonged QT syndrome, and use of medications that prolong QT
* Clinically serious thromboembolic disease within 6 months prior to the first administration of the study drug
* Major surgery within 4 weeks prior to the first administration
* History of severe gastrointestinal ulcers or perforations or history of intestinal obstruction within 6 months prior to the first administration
* Active infection requiring systemic treatment (oral or intravenous administration) within 2 weeks prior to the first administration, except for topical treatment
* History of non-infectious interstitial lung disease (ILD), such as idiopathic pulmonary fibrosis, idiopathic interstitial pneumonia, pneumoconiosis, and drug-related interstitial pneumonia, or severe impairment of lung function
* Had other malignancies within 5 years prior to screening (except clinically cured early stage malignancies)
* Primary central nervous system (CNS) tumor or symptomatic CNS metastasis, expect:

  * Subjects with asymptomatic brain metastases;
  * Subjects whose CNS lesions were stable for ≥4 weeks after local treatment and who stopped glucocorticoid or anticonvulsant therapy at least 2 weeks prior to study drug administration could be enrolled;
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Until 6 months after the last administration
  Incidence and severity of treatment emergent adverse events will be assessed as per CTCAE v5.0).
Dose-limiting toxicities (DLTs) during the DLT evaluation period | Up to 6 weeks after the first administration
  A DLT is defined as any drug-related toxicity that fulfills certain criteria predescribed in the study protocol.
Maximum tolerated dose (MTD) | Up to 6 weeks after the first administration
  MTD will be determined by 3+3 dose escalation design.
Recommended Phase 2 Dose (RP2D) | Through study completion, assessed up to 2 years
  RP2D will be determined on the basis of data indicating adequate tolerability and therapeutic effectiveness, and appropriate dosimestry. RP2D may be at or below the MTD.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Every 6 weeks after first administration until disease progression or through study completion, assessed up to 2 years
  ORR is defined as the proportion of participants with best overall response of Complete Response (CR) or Partial Response (PR) as measured by RECIST v1.1.
Duration of Response (DOR) | Every 6 weeks after first administration until disease progression or death or through study completion, assessed up to 2 years
  DOR is the time from the date of the first documented response (CR or PR) to the date of the first radiologically documented disease progression or death due to disease according to RECIST v1.1.
Disease Control Rate (DCR) | Every 6 weeks after first administration until disease progression or through study completion, assessed up to 2 years
  DCR is the percentage of participants with a best overall response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD) according to RECIST v1.1
Progression Free Survival (PFS) | Every 6 weeks after first administration until disease progression or death or through study completion, assessed up to 2 years
  PFS is defined as the interval from the date of first dosing to the date of first demonstrated disease progression, or to the last date of known progression-free condition of the patient, or to the date of death (based on RECIST 1.1).
Overall Survival (OS) | Every 6 weeks after first administration until death, assessed up to 2 years
  OS is defined as the interval from the date of first dosing to the date of death for any cause, or to the last date of known survival.
Radiation dosimetry of [177Lu]Lu-XT117 to whole body, lesions, organs, and selected regions of interest | 1、4、24、48、72 and 168 hours after first administration
  Radiation dosimetry is assessed by SPECT/CT and/or planar images.

CONTACTS AND LOCATIONS:
Overall Officials: Ruimin Wang, Principal Investigator — The First Medical Center, Chinese PLA General Hospital
Locations (1):
- The First Medical Center, Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu H, Guo R, Zhang X, Ji H, Sun S, Sun S, Liu J, Yang Z, Wang R. Safety and efficacy of 177Lu-FAPI-XT radioligand therapy in patients with advanced sarcoma and other cancer entities: first-in-human, dose-escalation study. Eur J Nucl Med Mol Imaging. 2025 Oct 15. doi: 10.1007/s00259-025-07617-0. Online ahead of print. PMID 41087606